CLINICAL TRIAL: NCT00279136
Title: Towards Restoring the Physiological Inhibition of Airway Narrowing in Asthma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: The Netherlands Asthma Foundation (Other)
Other Study IDs: AF 3.2.02.34, DIACON; Grant AF 3.2.02.34
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2006-01-19 (Estimated); Status verified 2005-09

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
Keywords: Bronchial hyperresponsiveness,; lung function,; airway inflammation,; deep inspiration,; bronchial biopsies; airway smooth muscle
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Bronchial Hyperreactivity

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Asthma and COPD are characterized by airway narrowing. The most potent, physiological mechanism leading to bronchodilation is taking a deep inspiration. This protects healthy subjects against bronchoconstrictive stimuli, and reverses pre-existing bronchoconstriction. However, the deep breath-induced bronchoprotection and -bronchodilation is impaired in asthma. We questioned whether this is specific for asthma (in comparison to COPD), and whether this is associated with bronchial inflammation and -remodelling. The study is a two-groups comparison, of physiological and pathological disease markers, obtained by methacholine challenges, monitoring airways resistance, and by taking bronchial biopsies.

DETAILED DESCRIPTION:
Rationale. Asthma is associated with variable airways obstruction and airways inflammation. It is generally assumed that inflammatory mechanisms are promoting airway narrowing, by stimulating airway smooth muscle and by geometrical changes of the airway wall. Healthy subjects are very effectively protected against stimuli of airway narrowing, by mechanisms that are apparently failing in asthma. The most potent inhibitor of airway narrowing in healthy subjects is taking a deep inspiration. This prevents and reverses bronchoconstriction (DI-induced bronchoprotection and -bronchodilation, respectively), which is less effective or absent in asthma. The DI-induced inhibition of airway narrowing in normal subjects is presumably due to relaxation of smooth muscle after mechanical stretch or to the release of relaxant mediators (such as endogenous NO). Such mechanisms might have become impaired in asthma, secondary to e.g. mechanical uncoupling of smooth muscle from the surrounding parenchyma (e.g. by congestion or edema), by altered structure and function of airway smooth muscle, and/or by reduced inhibitory mediator release.

It can be postulated that the impaired response to deep inspiration is a central pathophysiological feature of asthma at all ages. Therefore, we believe that it is imperative to address this, by identifying and restoring these inhibitory pathways in patients with asthma.

Hypotheses.

We hypothesize that DI-induced bronchoprotection and -broncho¬dilation:

1. are associated with cellular and morphological features of airways inflammation,
2. can be restored by deep insufflation rather than deep inspiration, and by pharmacological interventions aimed to reduce microvascular congestion or to increase endogenous nitric oxide synthesis..

Design and methods. To examine to what extent DI-responses differ between asthma and COPD in adulthood, and whether this is associated with features of airways inflammation and changes in smooth muscle function. 12 Adult patients with asthma and 12 with COPD will undergo single-dose methacholine challenge, with prohibition of DI's or 5 DI's prior to challenge in a cross-over design, measuring airways resistance. On a separate day bronchial biopsies will obtained with immunohistochemistry for inflammatory cell markers, vascularity, microvascular leakage, myosin light chain kinase, NO-synthases, and arginase.

ELIGIBILITY:
Inclusion Criteria:

* Asthma according to GINA criteria (www.ginasthma.org)
* COPD according to GOLD criteria (www.goldcopd.org)

Exclusion Criteria:

* nonsmoking
* inhaled or oral steroid therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2004-09; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Sterk, MD, PhD, Study Chair — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Derived] Slats AM, Janssen K, van Schadewijk A, van der Plas DT, Schot R, van den Aardweg JG, de Jongste JC, Hiemstra PS, Mauad T, Rabe KF, Sterk PJ. Bronchial inflammation and airway responses to deep inspiration in asthma and chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2007 Jul 15;176(2):121-8. doi: 10.1164/rccm.200612-1814OC. Epub 2007 Mar 22. PMID 17379851
- See also: Leiden University Medical Center — http://www.lumc.nl